CLINICAL TRIAL: NCT00408057
Title: Quality Enhancement Research Initiative (QERI) in the Dyslipidemia Management Strategy Involving Ezetimibe With Statin in High Risk Patients Who Have Not Achieved Recommended LDL Targets
Brief Title: Guidelines Based Undertaking for Improvement in Dyslipidemia Related Events (GUIDE )
Acronym: GUIDE
Status: Completed | Type: Observational
Sponsor: Canadian Heart Research Centre (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry); Schering-Plough (Industry)
Responsible Party: Dr. Shaun Goodman, Co-Chair, CHRC, Canadian Heart Research Centre
Other Study IDs: CHRC 020
Record Dates: First submitted 2006-12-01; First posted 2006-12-06 (Estimated); Last update posted 2008-05-14 (Estimated); Status verified 2008-05

CONDITIONS: Cardiovascular Diseases
Keywords: lipid lowering; target achievement; Patients with established cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — no intervenion

SUMMARY:
This is a multi-center, open label observational study conducted over 26 weeks.

Approximately 2,500 high-risk patients with an elevated LDL-C level (> 2.5 mmol/L) will be enrolled. Patients meeting all inclusion criteria and having none of the exclusion criteria at Visit 1 (Screening) will be included in the study. Eligible patients that agree to participate and sign an informed consent will be treated with either statin therapy (increased or started or switched) or combination of statin and ezetimibe 10 mg (added/started) as per Study Schematic (Table 1) in order to achieve the recommended target of LDL<2.5 mmol/L and providing that this treatment is in the best interest of the patient.

After enrollment there are a total of three scheduled clinic visits. All patients will have vital signs measured as well as a brief physical examination performed at Visit 1 (Screening).

At Visit 2 (6 weeks) patients with LDL-C > 2.5mmol/L will be treated with either statin therapy increase or combination of statin and ezetimibe 10 mg (added/started) as per Study Schematic (Table 1) in order to achieve the recommended target of LDL<2.5 mmol/L and providing that this treatment is in the best interest of the patient.

At Visit 3 (12 -18 weeks) patients with LDL > 2.5 mmol/L will be treated with combination of statin and ezetimibe 10 mg as per Study Schematic (Table 1) in order to achieve the recommended target of LDL<2.5 mmol/L and providing that this treatment is in the best interest of the patient.

At final Visit 4 (24-26 weeks) safety and efficacy of treatment will be reviewed. Following Visit 4 physicians will continue to treat these patients according to their clinical judgment.

DETAILED DESCRIPTION:
Overview This is a Quality Enhancement Research Initiative (QERI) whereby physicians are provided guidelines and easy to follow steps for their achievement..

Approximately 2,500 high-risk patients with an elevated LDL-C level (> 2.5 mmol/L) will be enrolled. Patients meeting all inclusion criteria and having none of the exclusion criteria at Visit 1 (Screening) will be included. Eligible patients that agree to participate and sign an informed consent will be treated with appropriate treatment optimization including the use of ezetimibe on achieving Study Schematics (Table 1).

After enrollment there are a total of three scheduled clinic visits. Physicians may assess the patient between visit 2 and 3 if maximization of statin therapy is required.

At Visit 2 (6 weeks) patients with LDL > 2.5mmol/L will be treated with either statin therapy (increased or started or switched) or combination of statin and ezetimibe 10 mg (added/started) as per Study Schematic (Table 1) in order to achieve the recommended target of LDL<2.5 mmol/L and providing that this treatment is in the best interest of the patient.

At Visit 3 (12-18 weeks) patients with LDL > 2.5 mmol/L will be treated with combination of statin and ezetimibe 10 mg (added/started) as per Study Schematic (Table 1) in order to achieve the recommended target of LDL<2.5 mmol/L and providing that this treatment is in the best interest of the patient.

At final Visit 4 (24-26 weeks) safety and efficacy of treatment will be reviewed. Following Visit 4 physicians will continue to treat these patients according to their clinical judgment.

1.5.1 Treatment

During this observational study patients will be treated under standard care with either statin therapy and/or co-administered with ezetimibe 10 mg /day. This is an open label observational study, therefore patients and physicians will be aware of treatment allocation and the treatment chosen will be that in the best interests of the patient and according to the physician's preference. Treatment will begin at Visit 1- Screening/Baseline (Day 0) and will extend through Visit 4 (Week 24-26).

Based on patient's LDL-C level, at visit 1 (Screening/Baseline) patient will receive prescription of initial or increased dose of statin 10-80 mg/day and/or ezetimibe 10 mg/day for the following 6 weeks. At visit 2 (6 weeks F/U) patients will receive prescription of statin (dose increased) and/or ezetimibe 10 mg per day for the following 6 weeks based on their target level of LDL-C. At visit 3 (week 12 -18 F/U) for patients who did not reach their LDL-C target, ezetimibe 10 mg per day will be considered if appropriate for the patient for the following 14 weeks to complete the observational study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female older 18 years of age.
2. Patients with a diagnosis of primary hypercholesterolemia and who are defined as being "high risk" (10-year risk of coronary artery disease greater than 20 % based on the Framingham model and history of cardiovascular disease or)
3. Patients who have not reached their recommended LDL-C target levels of 2.5 mmol/L while on a statin alone.
4. According to the judgment of the treating physician patient enrollment is in the best interest of the patient.
5. Patient agrees to participate and signs an informed consent allowing follow up and sharing of patient related data.

Exclusion Criteria:

1. Individuals with poor mental function, drug or substance abuse, or individuals with unstable psychiatric illnesses, which, in the opinion of the investigator, may interfere with optimal participation in the observational study. Alcoholic substance abuse would be defined as a patient with alcohol consumption > 14 drink per week. (A drink is: a can of beer, glass of wine, or single measure of spirits.)
2. Patients who have been treated with any investigational drug within 30 days prior to Visit 1. (If <30 days, contact the clinical monitor for a case-by-case evaluation.)
3. Patients with clinically significant concomitant illnesses of liver, muscle or kidney abnormalities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients considered at high risk for cardiovascular events
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2005-12; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Leiter, MD, Principal Investigator — University of Toronto
Locations (1):
- St. MIchael's Hospital, Toronto, Ontario, Canada